CLINICAL TRIAL: NCT05792904
Title: Factors Associated With Complicated Pneumonia in Paedatrics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marim Sedky Sedeek Ali, Factors associated with complicated pneumonia in paedatrics, Assiut University
Other Study IDs: Complicated pneumonia
Record Dates: First submitted 2023-03-17; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Complicated Pneumonia in Pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detecting Factors associated with complicated pneumonia in pediatrics

DETAILED DESCRIPTION:
Community acquired pneumonia is the cause of morbidity and mortality in children worldwide ,complication of Community acquired pneumonia in paedatrics include para -pneumonic pleural effusion ,empyema, necrotizing pneumonia and lung abscess.( Sawicki GS,2008) Pediatric para-pneumonic pleural effusion and empyema are considered different stages of the same pathophysiological process in which pleural inflammation causes fluid to accumulate in the pleural cavity, Necrotizing pneumonia results from pulmonary necrosis and tissue liquefaction. ( Ira Erlichman, MD,2017) Recent reports have characterized the clinical presentation of this complication and have shown favorable outcomes in children.( Sawicki GS,2008) Complicated pneumonia was defined as clinical pneumonia and the presence of pleural effusion, empyema (EMP) or Para-pneumonic childhood EMP was defined as the presence of pus (purulent fluid and/or WBC count>5,000 permm3) or bacteria in the pleural fluid.

PPE was defined by pleural fluid not fitting criteria of EMP and the diagnosis of NP was made by the presence of multiple cavity gas-filled spaces within a pulmonary consolidation on chest X-rays or liquefaction of lung tissue according to CT scans as reviewed by a pediatric radiologist .( Ira Erlichman, MD 2017) Among patients with pneumonia AS MANY AS half may develop pleural effusions (i.e., fluid in THE PLEURAL SPACE); of these, 5-10 % MAY DEVELOP EMPYEMAN Ingeneral , "complicated pneumonia" refers to pneumonia accompanied by pleural effusion.( Byington CL,2010) Empyema is a serious COMPLICATIO characterized by pus and bacteria in the pleural space which may progress to necrosis, cavitation, or fistulas in the thoracic cavity. S. pneumoniae is the most common cause of complicated pneumonia in children (an M. A. Fletcher ETT 2014) Empyema among children age below 19 years in Utah (USA) (1994-2007)] and Australia(1998-2010)ranged from 0.9 to 12.5 per 100,000 (Byington CL,2010)the incidence was highest in children aged 0-4 and tend to increase over time. (Strachan RE,2013).

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted at AUCH aged 2months up to 16 years old with sign and synptoms suggestive of pneumonia.

Exclusion Criteria:

* Immunodefiecency
* Hematological And Malignancy.
* NEONATAL PEROID.

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients included in the study will be divided into 3 groups Group1:patient with un complicated pneumonia. Group 2:patient who arrived with complicated pneumonia. Group3:patient who deveLoped pneumonia at hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
patients will be assessed by complete blood count | Baseline
C-reactive protein level | Baseline
Chest x-ray or CT chest image | Baseline

REFERENCES:
- [Result] McIntosh K. Community-acquired pneumonia in children. N Engl J Med. 2002 Feb 7;346(6):429-37. doi: 10.1056/NEJMra011994. No abstract available. PMID 11832532
- [Result] Sawicki GS, Lu FL, Valim C, Cleveland RH, Colin AA. Necrotising pneumonia is an increasingly detected complication of pneumonia in children. Eur Respir J. 2008 Jun;31(6):1285-91. doi: 10.1183/09031936.00099807. Epub 2008 Jan 23. PMID 18216055
- [Result] Sahn SA. Diagnosis and management of parapneumonic effusions and empyema. Clin Infect Dis. 2007 Dec 1;45(11):1480-6. doi: 10.1086/522996. Epub 2007 Oct 24. PMID 17990232
- [Result] Strachan RE, Snelling TL, Jaffe A. Increased paediatric hospitalizations for empyema in Australia after introduction of the 7-valent pneumococcal conjugate vaccine. Bull World Health Organ. 2013 Mar 1;91(3):167-73. doi: 10.2471/BLT.12.109231. Epub 2012 Dec 11. PMID 23476089